CLINICAL TRIAL: NCT06187454
Title: Transcranial Direct Current Stimulation for Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, Mu-N Liu, Principal Investigator, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-07-020B
Record Dates: First submitted 2023-11-21; First posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Experimental)
  Interventions: Device: Active Transcranial direct current stimulation
- Sham tDCS (Sham Comparator)
  Interventions: Device: Sham Transcranial direct current stimulation

INTERVENTIONS:
Device: Active Transcranial direct current stimulation — Transcranial direct current stimulation (tDCS) is a method for noninvasive brain stimulation, where a weak electrical current is delivered through two scalp electrodes by a portable battery-powered stimulator.
  Arms: Active tDCS
Device: Sham Transcranial direct current stimulation — For sham tDCS, the electrode positions and stimulation parameters will be the same as that used for anodal stimulation except that the current will be delivered only for the initial 30 seconds.
  Arms: Sham tDCS

SUMMARY:
Several studies have shown that tDCS is valuable and safe options to improve depressive symptoms in adult patients . However, regarding the tDCS to treat depression in elderly population, only few studies have been reported, and there is no consensus among them. To our knowledge, prefrontal cortex tDCS could be reasonably safe and efficient options for the treatment of several psychiatric illnesses in a population presenting resistance to and/or intolerance of pharmacotherapy . Moreover, the safety tolerability profile of tDCS is a strong argument in favour of exploring their use in the depressed population. Therefore, current study will investigate the efficacy and safety of prefrontal tDCS used as additive treatment in patients with LLD.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who meet the criteria of major depression defined by DSM-5 criteria
2. Participants will be non-responders and taking an antidepressant of adequate dose and for ≥4 weeks in the current episode which has not led to sufficient clinical improvement (defined as a minimum level of 2 on the ATHF); or can't tolerate the adverse effects of antidepressant in the current episode
3. Ambulatory participants with or without any aiding device

Exclusion Criteria:

1. An urgent risk of suicide or severe depression
2. A history of ineffectiveness with tDCS
3. People who are clinically contraindicated to receive tDCS intervention or MRI assessment, such as having any brain lesion, intracranial implants (clips, cochlear implants), a tattoo or metal embedded in their scalp or brain
4. Any instable medical condition
5. A history of epilepsy,
6. A history of substance use (within one year)
7. People with dementia or psychotic disorder.
8. Any condition which would make the subject unsuitable for the study under the physician's assessment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy and safety of tDCS | 8 Weeks
  [Primary Outcome Measures]
  * Hamilton Depression Rating Scale (HAMD) for depression
  * Comparison of these changes in both sham and active tDCS groups.
  * Response was defined as ≥ 50% HAMD score improvement from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- TaipeiVGH, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No